CLINICAL TRIAL: NCT00007579
Title: Prostate Cancer Case-Control Study: Black Versus White: VA Versus Private Sector
Brief Title: To Explore Racial Differences in Potential Risk Factors for Developing Prostate Cancer in the VA Population.
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Walther, Philip - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 708D
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2003-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Primary Objectives: To explore racial differences in potential risk factors for developing prostate cancer in the VA population and to compare and contrast the results of this study with that of an ongoing NCI-funded study in North Carolina.

Secondary Objectives: To investigate familial aggregation of prostate cancer in blacks and whites. To determine whether screening behavior differs in men diagnosed with early stage prostate cancer versus those with later stage disease as well as to determine if screening behavior differences exist between blacks and whites.

Primary Outcomes: The primary outcomes are pesticide, occupational and chemical exposure, and dietary history. Other major endpoints include: 1) familial aggregation of prostate cancer; 2) weight, weight history, and weight cycling; 3) subject's knowledge, attitudes, and behaviors about prostate cancer; and 4) treatment choices.

Intervention: N/A

Study Abstract: Prostate cancer is the most commonly diagnosed cancer in American men. Among African Americans the incidence and mortality from prostate cancer is even greater. Although incidence rates in the Southern United States tend to be only slightly higher than that of the nation, a clear discrepancy exists between national mortality rates and those in the Southeastern United States. Notably high rates, particularly among African Americans are observed and in North Carolina the prostate cancer mortality rate among African Americans is the highest of any state in the nation. In spite of these statistics, very little is known about racially based differences in the etiology of this disease.

This study hypothesizes that racial differences in the incidence and mortality of prostate cancer may be a result of multiple factors including those that are socioeconomic, environmental, dietary and genetic. This research will provide insight into gene-environmental interactions that initiate and promote prostatic neoplasia as well as address whether there are differences in patterns of care which impact morbidity and survival. The results of this study will also be compared to findings in non-veterans that are being generated through an NCI-funded sister study of these issues under the direction of co-investigator, Dr. JoEllen Schildkraut of Duke University.

Subjects were identified from pathology reports extracted from VISTA. Additionally, subjects were identified by reviewing radiation/oncology clinic records for those subjects referred for radiation treatment. Subject enrollment concluded with 100 cases and 98 controls enrolled in the study

DETAILED DESCRIPTION:
Primary Objectives: To explore racial differences in potential risk factors for developing prostate cancer in the VA population and to compare and contrast the results of this study with that of an ongoing NCI-funded study in North Carolina.

Secondary Objectives: To investigate familial aggregation of prostate cancer in blacks and whites. To determine whether screening behavior differs in men diagnosed with early stage prostate cancer versus those with later stage disease as well as to determine if screening behavior differences exist between blacks and whites.

Primary Outcomes: The primary outcomes are pesticide, occupational and chemical exposure, and dietary history. Other major endpoints include: 1) familial aggregation of prostate cancer; 2) weight, weight history, and weight cycling; 3) subject's knowledge, attitudes, and behaviors about prostate cancer; and 4) treatment choices.

Intervention: N/A

Study Abstract: Prostate cancer is the most commonly diagnosed cancer in American men. Among African Americans the incidence and mortality from prostate cancer is even greater. Although incidence rates in the Southern United States tend to be only slightly higher than that of the nation, a clear discrepancy exists between national mortality rates and those in the Southeastern United States. Notably high rates, particularly among African Americans are observed and in North Carolina the prostate cancer mortality rate among African Americans is the highest of any state in the nation. In spite of these statistics, very little is known about racially based differences in the etiology of this disease.

This study hypothesizes that racial differences in the incidence and mortality of prostate cancer may be a result of multiple factors including those that are socioeconomic, environmental, dietary and genetic. This research will provide insight into gene-environmental interactions that initiate and promote prostatic neoplasia as well as address whether there are differences in patterns of care which impact morbidity and survival. The results of this study will also be compared to findings in non-veterans that are being generated through an NCI-funded sister study of these issues under the direction of co-investigator, Dr. JoEllen Schildkraut of Duke University.

Subjects are identified from pathology reports extracted from VISTA. It has been determined that pathology reports alone are not a sufficient source of identifying cases because not all patients coming to VA for treatment have diagnostic pathology completed at the Durham VA. Therefore, we have added additional protocols for subject identification such as reviewing radiation/oncology clinic records for those subjects referred for radiation treatment. To-date, 78 cases and 66 controls have been enrolled in the study. To increase accrual rates, in-home visits have been used when necessary, and the Richmond, VA and Asheville, NC VAMCs have been added as participating study sites. Due to patient accrual problems and project staffing changes, the Durham ERIC has granted this study a six-month, no-cost extension through 7/31/2001.

ELIGIBILITY:
Inclusion Criteria:

Veterans with Prostate Cancer

Exclusion Criteria:

Ages: 40 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-02

CONTACTS AND LOCATIONS:
Overall Officials: Philip Walther, Study Chair — VA Medical Center, Durham
Locations (1):
- VA Medical Center, Durham, Durham, North Carolina, United States